CLINICAL TRIAL: NCT05946200
Title: Comparison of the Effects of Low-flow and Normal-flow on Intracranial Pressure, Cerebral Oxygenation, and Bispectral Index in Laparoscopic Cholecystectomy Operation
Brief Title: Optic Nerve Sheath Diameter in Low-flow and Normal-flow Rate Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Aydın Mermer, Vice Director, Head of Anesthesiology, Principal Investigator, Clinical Specialistsor, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023/4146 (12662)
Record Dates: First submitted 2023-06-02; First posted 2023-07-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Intracranial Hypertension
Keywords: Low flow anesthesia; optic sheath diameter; intracranial pressure; laparoscopic cholecystectomy
MeSH Terms: conditions — Intracranial Hypertension | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the care provider will know what's going on in the management of the patient. Cause that they should manage the case properly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low flow (Active Comparator): It will be used low-flow (0.75 l/min) to manage the general anesthesia.
  Interventions: Procedure: Low flow technique in general anesthesia
- Normal flow (Sham Comparator): It will be used normal-flow (1.5 l/min) to manage the general anesthesia.
  Interventions: Procedure: Low flow technique in general anesthesia

INTERVENTIONS:
Procedure: Low flow technique in general anesthesia — It will be used a low flow technique by giving airflow as 0.75 l/min after the intubation and will keep going on until the end of the laparoscopic cholecystectomy.

SUMMARY:
Laparoscopic cholecystectomy is one of the regularly performed laparoscopic surgical procedures. It resulted in shorter hospital stays, improved cosmetic outcomes, and reduced bleeding and pain. However, during laparoscopic surgeries, the pneumoperitoneum is known to raise intracranial pressure (ICP), reduction in cerebral blood flow (CBF), and as a consequence, cerebral hypoxia. There are various possible advantages of low-flow anesthesia. During laparoscopic procedures, low-flow anesthesia may be used as a means of preventing a rise in intracranial pressure and cerebral hypoxia. But low flow anesthesia effects on İCP are not known in Laparoscopic cholecystectomy. The primary aim of this study is to compare the effects of low-flow (0.75 l/min) and normal-flow (1.5 l/min) anesthesia on ONSD in patients undergoing laparoscopic cholecystectomy. Seconder aims are regional cerebral oxygen saturation (rSO2), bispectral index (BIS), and evaluate the status of cognitive function in the postoperative 24th hours.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the regularly performed laparoscopic surgical procedures. It resulted in shorter hospital stays, improved cosmetic outcomes, and reduced bleeding and pain. However, during laparoscopic surgeries, the pneumoperitoneum is known to raise intracranial pressure (ICP), reduction in cerebral blood flow (CBF), and as a consequence, cerebral hypoxia.

Near-infrared spectroscopy (NIRS), a noninvasive and continuous measuring method used to evaluate the appropriateness of cerebral perfusion, is therefore utilized in conjunction with cerebral oximetry to quantify regional tissue oxygenation. On the other, BIS is the most reliable technique for determining the level of sedation and anesthesia. Patients experience fewer intraoperative wake-ups thanks to BIS monitoring. Increased intra-abdominal pressure, decreased cerebrospinal fluid (CSF) absorption and obstruction of lumbar venous plexus drainage, increased pressure in the sacral spaces' vascular compartment, and cerebral vasodilation brought on by hypercarbia are some of the suggested mechanisms for why ICP increases during laparoscopy. Intraventricular and intraparenchymal catheterization remains the gold standard for determining and monitoring ICP. However, due to worries about severe complications like bleeding, infection, and equipment failure, invasive ICP monitoring during laparoscopic surgery is almost impossible. Recently, ultrasound-guided optic nerve sheath diameter (ONSD) measurement is a simple and reliable method of predicting elevated ICP.

There are various possible advantages of low-flow anesthesia. It boosts mucociliary clearance, preserves body temperature, lessens fluid loss, generates savings of up to 75%, and lowers greenhouse gas emissions as well as the cost of treatment. It also improves the flow dynamics of the breathed air. During laparoscopic procedures, low-flow anesthesia may be used as a means of preventing a rise in intracranial pressure and cerebral hypoxia. But low flow anesthesia effects on İCP are not known in Laparoscopic cholecystectomy.

The primary aim of this study is to compare the effects of low-flow (0.75 l/min) and normal-flow (1.5 l/min) anesthesia on ONSD in patients undergoing laparoscopic cholecystectomy. Seconder aims are regional cerebral oxygen saturation (rSO2), bispectral index (BIS), and evaluate the status of cognitive function in the postoperative 24th hours.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria of the patients will be determined as age between 18 and 65 years, ASA status 1-2.

Exclusion Criteria:

* Exclusion criteria of the patients are defined as patients younger than 18, pregnant women, patients with any ophthalmological disease affecting optic nerve diameters, patients with acute or chronic eye disease, patients using drugs known to affect intracranial pressure, and patients abusing alcohol or psychoactive substances.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter. | Intraoperative period
  The primer outcome of this study is to measure optic nerve sheath diameter during by using low-flow (0.75 l/min) and normal-flow (1.5 l/min) anesthesia on ONSD in patients undergoing laparoscopic cholecystectomy.

SECONDARY OUTCOMES:
Regional cerebral oxygen saturation (rSO2) | Intraoperative period
  Seconder outcome 1 is regional cerebral oxygen saturation (rSO2) between low and normal flow technique.
Bispectral index (BIS) | Intraoperative period
  Seconder outcome 2 is bispectral index (BIS) between low and normal flow technique.
Cognitive function assessment by using Mini mental test | Perioperative period.
  Seconder aim 3 is to get Mini mental test score in the postoperative 24th.hours.

CONTACTS AND LOCATIONS:
Overall Officials: Aydın Mermer, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No